CLINICAL TRIAL: NCT04722029
Title: Open-Label Pilot Study of Haploidentical Donor Adenovirus Specific T Lymphocytes (ADV-VSTS) for the Treatment of Refractory Adenovirus Infection and/or Disease in Hospitalized Patients
Brief Title: Pilot Study of Haploidentical Donor Adenovirus Specific T-lymphocytes to Treat Refractory Adenovirus Infections
Acronym: ADV-VSTS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001291
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Adenovirus Infection
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Donor (No Intervention): Donors will be evaluated to determine suitability to undergo apheresis collection and their infectious disease status. Donor evaluation will include history and physical examination, laboratory tests, FDA- approved donor testing of communicable diseases (HIV, HVB, HCV, HTLV-I, II, WNV, T. pallidum, T. cruzi, and Zika virus), ABO and Rh typing, pregnancy tests, and donor serology for ADV.
  Qualified donors will undergo leukapheresis. Collection will proceed for 2 hours or 2 blood volumes, whichever occurs first.
- Recipient (Experimental): Recipient will undergo a screening period that will include history and physical examination, laboratory tests, performance status, HLA typing and pregnancy test (if needed).
  Qualified patients will receive ADV-VSTS infusion from haploidentical donors up to a maximum of 5.0 x 104 interferon gamma-negative cells/kg. All patients will be followed for laboratory and clinical response, safety, efficacy and tolerance.
  Interventions: Biological: Adenovirus Specific T lymphocytes

INTERVENTIONS:
Biological: Adenovirus Specific T lymphocytes — ADV-VSTs is being proposed for the treatment of refractory ADV infection and/or disease in these populations using haploidentical donors for ease of donor selection, antiviral immunity, coupled with a high-throughput antigen stimulation/IFN-γ capture system (Miltenyi Biotec, CliniMACS Prodigy® System) for rapid and less costly isolation of ADV-VSTs.
  Arms: Recipient

SUMMARY:
This open-label, single-arm, phase I/II clinical trial will assess the safety and efficacy of related donor adenovirus-specific T lymphocytes isolated from whole blood or leukapheresis products. The adenovirus-specific T lymphocytes will be generated automatically by the CliniMACS Prodigy using the CliniMACS Cytokine Capture System (IFN-γ) after incubation with MACS GMP PepTivator Peptide Pools of Hexon 5 for enrichment.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 days to 60 years with one of the following conditions:

  1. Patients who are solid organ transplantation recipients (renal, heart, lung, liver, pancreas, small bowel, multi-visceral) and are > 28 days post-transplant at the time of screening.
  2. Patients with underlying malignancy who are receiving or have received chemotherapy within 6 months of screening.
  3. Patients with known autoimmune or autoinflammatory conditions, not associated with a known underlying primary immunodeficiency
  4. Patients who are receiving or have received systemic immunosuppressive therapies in the 30 days prior to screening including: biologic agents, calcineurin inhibitors, mTOR inhibitors, or corticosteroid
  5. Patients without known immunocompromised conditions
* And must meet at least 1 of the following criteria.

  1. Documented ADV refractory infection (i.e., DNAemia detected by qualitative or quantitative PCR in the peripheral blood > 14 days or rising viral load in blood despite antiviral therapy >14 days).
  2. Evidence of refractory ADV end organ disease (proven or probable as previously defined46, including pneumonitis, colitis, hepatitis, hemorrhagic cystitis etc.) despite antiviral therapy >14 days.
  3. Medical intolerance to anti-viral therapies including renal toxicity (Cr >2) and/or bone marrow suppression (ANC <1500, Hb <10 and/or Plt <50) or gastrointestinal manifestation (grade ≥2 diarrhea), or other related organ injury.
  4. At high risk for antiviral failure due to history of recurrent ADV reactivations, or recently started on increased immunosuppressants.
* Negative pregnancy test in female patients if applicable (childbearing potential)
* Written informed consent and/or signed assent line from patient, parent or legal guardian prior to any study-related procedures.

Exclusion Criteria:

* Receipt of anti-thymocyte globulin (ATG), alemtuzumab, cytoxan, or other T-cell depleting drugs or monoclonal antibodies within 28 days from enrollment
* Receiving corticosteroid (prednisone equivalent) ≥ 0.5mg/kg/day or ≥ 20mg/day at the time of enrollment
* Recipients of allogeneic hematopoietic stem cell transplant (bone marrow, peripheral blood or umbilical cord blood)
* Evidence of uncontrolled infection (except ADV) as follows:

  1. Bacterial infections - patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment
  2. Fungal infections - patients must be receiving definitive systemic anti-fungal therapy and evidence of response/stabilization on therapy for 1 week prior to enrollment
  3. Progressing infection is defined as hemodynamic instability attributable to sepsis, or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection
* Patient with poor performance status determined by Karnofsky (patients >16 years) or Lansky (patients ≤16 years) score ≤30% (Table 5)
* Concomitant enrollment in another experimental clinical trial investigating the treatment of refractory adenovirus infection(s)
* During the study, treatment with other investigational anti-adenoviral agents is prohibited until Week 12.
* If patient has been treated with CMX001 (brincidofovir, BCV) prior to ADV-VST enrollment, BCV must be discontinued for at least 72 hours prior to ADV-VSTs infusion for washout based on known geometric mean elimination half-life of BCV (8 to 12 hours). Any medical condition which could compromise participation in the study according to the investigator's assessment
* Known HIV infection
* Female patient of childbearing age who is pregnant or breast-feeding or not willing to use an effective method of birth control during study treatment.
* Known hypersensitivity to iron dextran
* Patients unwilling or unable to comply with the protocol or unable to give informed consent.
* Known human anti-mouse antibodies

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety by measuring unacceptable toxicities | 7-28 days
  Safety will be assess at 28 days post ADV-VSTS infusion. Safety is defined as presentation of unacceptable toxicities, measured by grade III-IV acute GVHD within 28 days, solid organ rejection/ graft failure within 28 days, grade >4 infusional toxicity within 7 days of infusion, and grade 4-5 adverse events within 28 days per CTCAE 5.0.
Efficacy by measuring viral load | 28 days
  Percentage of patients with ≥1 log decrease in ADV viral load. ADV viral load will be monitored by quantitative ADV PCR weekly until negative PCR. Response will be assess on day 28 post ADV-VSTS infusion defined as complete response, partial response, stable disease or progressive disease

CONTACTS AND LOCATIONS:
Overall Officials: Eunkyung Song, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No